CLINICAL TRIAL: NCT00766415
Title: A Double-blind, Placebo-controlled, Randomised, Parallel Group Phase IIa Study to Evaluate the Histological Changes, Cellularity, Clinical Efficacy and Safety of AZD1981 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: 14729-D9831C00002- 1 Month Biopsy Study
Acronym: Biopsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9831C00002
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Moderate to severe COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — AZD1981

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD1981 (Experimental)
  Interventions: Drug: AZD1981
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1981 — Oral tablet, twice daily, 4 weeks treatment
  Arms: AZD1981
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to study histological changes, cellularity, clinical efficacy and safety of AZD1981 in patients with Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion Criteria:

* Men or women 40 years or above
* FEV1 between 40 and 80% of predicted normal value post-bronchodilator
* Clinical diagnosis of COPD

Exclusion Criteria:

* Other clinically relevant disease or disorders
* Exacerbation of COPD within 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-11; Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Krug, Principal Investigator — Fraunhofer Institute
Locations (8):
- Germany (3):
  - Research Site, Frieburg
  - Research Site, Großhansdorf
  - Research Site, Hanover
- Research Site, Amsterdam, Netherlands
- United Kingdom (4):
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=216&filename=CSR-D9831C00002.pdf
- See also: CSR-D9831C00002.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=216&filename=CSR-D9831C00002.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 patients enrolled, 52 were randomised, 1 patient discontinued before treatment start and 51 patients completed the study. First patient entered the study on 17 November 2008 and the last patient finished the study on 10 June 2009.
Groups:
- AZD1981: AZD1981 1000 mg, twice daily
- Placebo: Placebo, twice daily
Period: Overall Study
Arm/Group | AZD1981 | Placebo
Started | 25 | 27
Completed | 25 | 26
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient randomised to the placebo group voluntarily discontinued from the study after randomisation before receiving any investigational product. This patient is excluded from the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1981 | Placebo | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Full Range); unit: Years] — 1 participant discontinued immediately following randomization, did not start treatment and have not been included in any of the efficacy or safety calculations.
  Years | 61 [50 to 75] | 61.1 [41 to 80] | 61 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — 1 participant discontinued immediately following randomization, did not start treatment and have not been included in any of the efficacy or safety calculations.
  Participants
    Female | 9 | 4 | 13
    Male | 16 | 22 | 38

OUTCOME MEASURES:

1. Primary Outcome: Aggregated Pathology Score
Description: Composite endpoint subscores: histological grade, immunohistochemistry grade, leucocyte counts. Each subscore measured on scale 1 (normal) to 5 (worst outcome). Composite score summed across the subscores, ranging from 3 (normal) to 15 (worst outcome). Change from baseline.
Time Frame: Before and after 1 month treatment
Population: Efficacy analyses were performed on the full-analysis set, comprised of 51 patients: 25 in the AZD1981 group and 26 in the placebo group. However, not all patients will have valid, non-missing values for a given outcome measure.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 24 | 26
Score on a scale | 7.88 (7.43) [7.43 to 8.34] | 8.15 (7.68) [7.68 to 8.63]

2. Primary Outcome: Bronchoalveolar Lavage (BAL): Eosinophil Count (%)
Description: Change in Bronchoalveolar Lavage (BAL): Eosinophil count (% of total) from baseline
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 21 | 22
percentage | -1.58 (-2.22) [-2.22 to -0.94] | -1.45 (-2.13) [-2.13 to -0.78]

3. Primary Outcome: Bronchoalveolar Lavage (BAL): Neutrophil Count (%)
Description: Change in Bronchoalveolar Lavage (BAL): Neutrophil count (% of total) from baseline
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 21 | 22
percentage | -2.24 (-12.94) [-12.94 to 8.46] | -5.67 (-16.75) [-16.75 to 5.42]

4. Primary Outcome: Bronchoalveolar Lavage (BAL): Macrophages Count (%)
Description: Change in Bronchoalveolar Lavage (BAL): Macrophages count (% of total) from baseline
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 21 | 22
percentage | 9.84 (-1.51) [-1.51 to 21.20] | 10.68 (-1.24) [-1.24 to 22.60]

5. Primary Outcome: Bronchoalveolar Lavage (BAL): Lymphocytes Count (%)
Description: Change in Bronchoalveolar Lavage (BAL): Lymphocytes count (% of total) from baseline
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 21 | 22
percentage | -1.47 (-3.04) [-3.04 to 0.11] | -0.37 (-2.02) [-2.02 to 1.28]

6. Primary Outcome: Bronchoalveolar Lavage (BAL): Epithelial Cells Count (%)
Description: Change in Bronchoalveolar Lavage (BAL): Epithelial cells count (% of total) from baseline
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 21 | 22
percentage | -4.18 (-11.80) [-11.80 to 3.45] | -2.98 (-10.98) [-10.98 to 5.01]

7. Primary Outcome: Bronchoalveolar Lavage (BAL): Total Cells Count
Description: Change in Bronchoalveolar Lavage (BAL): Total cells count from baseline
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: 10^6/g
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 23 | 24
10^6/g | 0.02 (-0.10) [-0.10 to 0.15] | 0.04 (-0.10) [-0.10 to 0.17]

8. Primary Outcome: Induced Sputum: Eosinophil Count (%)
Description: Change in Induced sputum Eosinophil count (% of total) from baseline
Time Frame: Before and after 3 week treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 14 | 17
percentage | -2.14 (-3.30) [-3.30 to -0.98] | -0.81 (-1.92) [-1.92 to 0.30]

9. Primary Outcome: Induced Sputum: Neutrophils Count (%)
Description: Change in Induced sputum Neutrophils count (% of total) from baseline
Time Frame: Before and after 3 week treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 14 | 17
percentage | 0.70 (-12.79) [-12.79 to 14.19] | 3.73 (-8.84) [-8.84 to 16.30]

10. Primary Outcome: Induced Sputum: Macrophages Count (%)
Description: Change in Induced sputum Macrophages count (% of total) from baseline
Time Frame: Before and after 3 week treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 14 | 17
percentage | 1.31 (-11.95) [-11.95 to 14.57] | -7.79 (-20.27) [-20.27 to 4.69]

11. Primary Outcome: Induced Sputum: Lymphocytes Count (%)
Description: Change in Induced sputum Lymphocytes count (% of total) from baseline
Time Frame: Before and after 3 week treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 14 | 17
percentage | -0.01 (-0.21) [-0.21 to 0.18] | 0.02 (-0.17) [-0.17 to 0.20]

12. Primary Outcome: Induced Sputum: Epithelial Cells Count (%)
Description: Change in Induced sputum Epithelial cells count (% of total) from baseline
Time Frame: Before and after 3 week treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 14 | 17
percentage | -0.50 (-6.01) [-6.01 to 5.01] | 4.11 (-1.04) [-1.04 to 9.27]

13. Primary Outcome: Induced Sputum: Total Cells Count
Description: Change in Induced sputum Total cells count from baseline
Time Frame: Before and after 3 week treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: 10^6/g
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 19 | 17
10^6/g | -1.07 (-3.21) [-3.21 to 1.08] | -1.69 (-4.07) [-4.07 to 0.69]

14. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Change in Forced Expiratory Volume in 1 second (FEV1) from baseline to end of treatment
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 26
percentage change | -4.77 (-15.94) [-15.94 to 6.40] | 6.16 (-5.66) [-5.66 to 17.97]

15. Secondary Outcome: Clinical Chronic Obstructive Pulmonary Disease (COPD) The Clinical COPD Questionnaire (CCQ)
Description: Change in total CCQ score from baseline to last measurement on treatment. scored on a scale of 0 - 6. 0 =(low symptoms)-6 =(high symptoms)
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 24
Scores on a scale | -0.38 (-0.69) [-0.69 to -0.06] | -0.34 (-0.68) [-0.68 to 0.00]

16. Secondary Outcome: Peak Expiratory Flow (PEF) Morning
Description: Mean change in Peak Expiratory Flow (PEF) morning from baseline to the average of the treatment period
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 24
L/min | 2.57 (-9.55) [-9.55 to 14.69] | -4.14 (-16.96) [-16.96 to 8.69]

17. Secondary Outcome: Peak Expiratory Flow (PEF) Evening
Description: Mean change in Peak Expiratory Flow (PEF) evening from baseline to the average of the treatment period
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 21
L/min | 1.31 (-13.03) [-13.03 to 15.65] | 1.46 (-14.27) [-14.27 to 17.19]

18. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Symptom Night-time Awakenings Score
Description: Mean change in COPD symptom night-time awakening score from baseline to the average of the treatment period. 0=(no symptom)-4=(no sleep)
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 24
Score on a scale | -0.23 (-0.47) [-0.47 to 0.01] | -0.24 (-0.49) [-0.49 to 0.02]

19. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Symptom Breathing Score
Description: Mean change in COPD symptom breathing score from baseline to the average of the treatment period. 0= (none) - 4 =(severe).
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 21
Score on a scale | -0.25 (-0.47) [-0.47 to -0.03] | -0.21 (-0.45) [-0.45 to 0.04]

20. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Symptom Cough Score
Description: Mean change in COPD symptom cough score from baseline to the average of the treatment period. 0= (none) - 4= (almost constant)
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 21
Score on a scale | -0.39 (-0.63) [-0.63 to -0.16] | -0.35 (-0.61) [-0.61 to -0.09]

21. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Symptom Sputum Score
Description: Mean change in COPD symptom sputum score from baseline to the average of the treatment period. 0= (none) - 4= (severe).
Time Frame: Before and after 1 month treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 21
Score on a scale | -0.32 (-0.52) [-0.52 to -0.12] | -0.38 (-0.60) [-0.60 to -0.16]

22. Secondary Outcome: Adverse Event (AE)
Description: Number of participants with an Adverse Event
Time Frame: 1 month
Measure: Number; unit: Participants
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 25 | 26
Participants | 17 | 14

ADVERSE EVENTS:
Description: 1 participant discontinued immediately following randomization, did not start treatment and have not been included in any of the efficacy or safety calculations.
Arm/Group | AZD1981 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/26
Other Adverse Events (participants affected / at risk) | 5/25 | 7/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 (N=25) | Placebo (N=26)
Hypoxia After Bronchoscopy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 (N=25) | Placebo (N=26)
Nasopharyngitis (Infections and infestations) | 3 | 2
Headache (Nervous system disorders) | 1 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less